CLINICAL TRIAL: NCT05180695
Title: A Multicenter, Phase I/II Study Evaluating the Clinical Impact of HDM201 + Pazopanib in Patients With P53 Wild-type Advanced/ Metastatic Soft Tissue Sarcomas (AMPHISARC)
Brief Title: HDM201 and Pazopanib in Patients With P53 Wild-type Advanced/Metastatic Soft Tissue Sarcomas
Acronym: AMPHISARC
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: Novartis (Industry); National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ET20-297
Record Dates: First submitted 2021-12-07; First posted 2022-01-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Advanced Soft-tissue Sarcoma; Metastatic Soft-tissue Sarcoma
Keywords: P53 wild type; pazopanib; HDM201; RECIST
MeSH Terms: conditions — Sarcoma | interventions — pazopanib; siremadlin

STUDY DESIGN:
Intervention Model Description: The dose escalation will be conducted according to a sequential and adaptive Bayesian scheme, using the method of TITE-CRM to determine the MTD of pazopanib in combination with HDM201. This method allows continual accrual (i.e. the study will be opened to accrual continually) throughout the trial while using the 6-week toxicity endpoint as basis of dose escalation.
  Dose allocation will be centrally defined, before each inclusion considering the DLT observed in all patients previously evaluated, and the current toxicity status of patients who have not received a full 2-cycle treatment (i.e. DLT period is still ongoing).
  * A cumulative experience of 4 cycles at a given DL is required before allowing dose escalation to the next DL. Cumulative experience is defined as the addition of observation periods of all included and treated patients.
  * A maximum of 6 patients can be included and treated at a same dose level before reassessment occurred.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- extension part : Soft-tissue sarcomas with MDM2 amplification (Experimental): The aim of each extension cohort is to provide preliminary evidence of anti-tumor activity while refining toxicity data, and to gain insight progressive disease activity and exploratory biological analyses. A maximum of 14 patients patients will be enrolled in this cohort " Soft-tissue sarcomas with MDM2 amplification ". Both study drugs (pazopanib and HDM201) will be administered as long as the patient experiences clinical benefit in the opinion of the investigator or until unacceptable toxicity or symptomatic deterioration attributed to disease progression as determined by the investigator after an integrated assessment of radiographic data and clinical status or withdrawal of consent.
  Interventions: Drug: Pazopanib; Drug: HDM201
- extension part : Soft-tissue sarcomas with no MDM2 amplification (Experimental): A maximum of 14 patients patients will be enrolled in this cohort " Soft-tissue sarcomas with no MDM2 amplification". Both study drugs (pazopanib and HDM201) will be administered as long as the patient experiences clinical benefit in the opinion of the investigator or until unacceptable toxicity or symptomatic deterioration attributed to disease progression as determined by the investigator after an integrated assessment of radiographic data and clinical status or withdrawal of consent.
  Interventions: Drug: Pazopanib; Drug: HDM201

INTERVENTIONS:
Drug: Pazopanib — Part 1: A dose escalation part with the aim to assess the safety of the proposed combination. Eligible patients will be treated with a fixed dose of pazopanib (800mg/d, continuously) and escalating doses of HDM201. Both study drugs will be administered as long as the patient experiences clinical benefit in the opinion of the investigator or until unacceptable toxicity or symptomatic deterioration attributed to disease progression or withdrawal of consent.
  Part 2: An extension part with a fixed dose of pazopanib (800mg/d, continuously) and the recommended phase 2 dose of HDM201 determined during the dose escalation part. Both study drugs will be administered as long as the patient experiences clinical benefit in the opinion of the investigator or until unacceptable toxicity or symptomatic deterioration attributed to disease progression or withdrawal of consent.
  Other Names: Votrient
Drug: HDM201 — Part 1: A dose escalation part with the aim to assess the safety of the proposed combination. Eligible patients will be treated with a fixed dose of pazopanib (800mg/d, continuously) and escalating doses of HDM201. Both study drugs will be administered as long as the patient experiences clinical benefit in the opinion of the investigator or until unacceptable toxicity or symptomatic deterioration attributed to disease progression or withdrawal of consent.
  Part 2: An extension part with a fixed dose of pazopanib (800mg/d, continuously) and the recommended phase 2 dose of HDM201 determined during the dose escalation part. Both study drugs will be administered as long as the patient experiences clinical benefit in the opinion of the investigator or until unacceptable toxicity or symptomatic deterioration attributed to disease progression or withdrawal of consent.
  Other Names: siremadlin

SUMMARY:
This trial is a two-step Phase I/II study comprising:

Part 1: A dose escalation part with the aim to assess the safety of the proposed combination (N= up to 30 patients). In the dose escalation part, eligible patients will be treated with a fixed dose of pazopanib and escalating doses of HDM201.

Part 2: An extension part to collect preliminary data about the clinical activity of the proposed combination according to the 6M-PFR.

DETAILED DESCRIPTION:
This trial is a two-step Phase I/II study comprising:

Part 1: A dose escalation part with the aim to assess the safety of the proposed combination (N= up to 30 patients). The dose escalation will be conducted according to a sequential and adaptive Bayesian scheme using the method of Time-to-event Continual Reassessment Method (CRM) to guide dose escalation and estimate the Maximum Tolerated Dose.

In the dose escalation part, eligible patients will be treated with a fixed dose of pazopanib (800 mg/d) and escalating doses of HDM201: 60 mg (starting dose); 80 mg; 100 mg; 120 mg. For a safety reason, a dose level of 40 mg is included in case that the first dose level is found to be toxic. In addition, decrease of pazopanib dosing to 600 mg/d could be appropriate following protocol amendment.

To ensure adequate patient safety during the dose escalation part, there will be a 3-day delay between the first and subsequent patients enrolled in each DL cohort to maximize the safety of enrolled patients.

No intra-patient dose escalation is allowed.

Part 2: An extension part to collect preliminary data about the clinical activity of the proposed combination according to the 6 months Progression Free Rate (6M-PFR).

ELIGIBILITY:
Inclusion Criteria:

I1. Male or female patient ≥ 18 years of age

I2. Histologically or cytologically confirmed diagnosis of soft tissue sarcoma with documented p53 wild-type (wt) status and known MDM2 status (amplification or no amplification).

Note: p53 wt status has to be determined by Next-generation sequencing of the full coding sequence using a tumor sample collected no longer than 36 months before inclusion.

I3. Previously treated by at least one prior chemotherapy line of treatment in the advanced/metastatic setting.

I4. STS subtypes eligible to pazopanib treatment according to respective SmPC Note: The following tumour types are eligible: Fibroblastic (adult fibrosarcoma, myxofibrosarcoma, sclerosing epithelioid fibrosarcoma, malignant solitary fibrous tumours), so-called fibrohistiocytic (pleomorphic malignant fibrous histiocytoma [MFH], giant cell MFH, inflammatory MFH), leiomyosarcoma, malignant glomus tumours, skeletal muscles (pleomorphic and alveolar rhabdomyosarcoma), vascular (epithelioid hemangioendothelioma, angiosarcoma), uncertain differentiation (synovial, epithelioid, alveolar soft part, clear cell, desmoplastic small round cell, extra-renal rhabdoid, malignant mesenchymoma, PEComa, intimal sarcoma), malignant peripheral nerve sheath tumours, undifferentiated soft tissue sarcomas not otherwise specified (NOS) and other types of sarcoma (not listed as ineligible)and liposarcoma.

The following tumour types ARE NOT eligible: All rhabdomyosarcoma that are not alveolar or pleomorphic, chondrosarcoma, osteosarcoma, Ewing tumours/primitive neuroectodermal tumours (PNET), GIST, dermofibromatosis sarcoma protuberans, inflammatory myofibroblastic sarcoma, malignant mesothelioma and mixed mesodermal tumours of the uterus

I5. Documented progressive disease and presence of at least one measurable lesion according to RECIST 1.1 (Appendix 01) based on screening tumor assessment.

I6. Performance Status score of 0 or 1 according to the Eastern Cooperative Oncology Group (ECOG) scale.

I7. Adequate organ system function as assessed by the following minimal requirements (within 7 days prior to first administration of study drugs (C1D1)):

Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L Platelets ≥ 100 x 109/L Hemoglobin ≥ 9 g/dL (5.6 mmol/L). Transfusion is not allowed within 2 weeks of screening assessment.

aspartate transaminase and alanine aminotransferase ≤ 2.5x Upper limit of normal or up to 5 Upper limit of normal in case of liver metastasis Bilirubin ≤ 1.5 Upper limit of normal (except in the setting of isolated Gilbert syndrome) Serum creatinine clearance ≥ 30 mL/min (calculated by CKD-EPI -Appendix 03) Calcium, magnesium and potassium within normal limits. Urine Protein to Creatinine ratio (UPC) <1; if UPC ≥1, 24-hour urine protein must be <1g (use of urine dipstick for renal function assessment is not acceptable).

I8. Adequate cardiovascular function:

QTcF (corrected QT using Fridericia) ≤450ms, from 3 electrocardiograms on screening ECG, within 14 days prior to C1D1 Resting blood pressure systolic <140 mmHg and diastolic< 90 mmHg, Left Ventricular Ejection Fraction ≥50% as determined by transthoracic echocardiogram or Multiple Gated acquisition.

I9. Resolution (i.e. ≤ Grade 1 with the exception of alopecia all grades and Grade 2 for neuropathy, lab values presented in inclusion criteria) of any toxicities related to previous anti-cancer treatment.

I10. Patients able to swallow orally administered medication and do not have any clinically significant gastrointestinal abnormalities that may alter absorption of study drugs such as malabsorption syndrome or major resection of the stomach or bowels.

I11. Availability of archival Formalin Fixed Paraffin Embedded tumor sample. This sample must be sent to sponsor once eligibility is confirmed.

I12. Expansion part only - Presence of at least one biopsiable lesion i.e. at least one lesion with a diameter ≥10 mm, visible by medical imaging and accessible to repeatable percutaneous or endoscopic sampling that permit core needle biopsy without unacceptable risk and suitable for retrieval of a minimum of three, but ideally four, cores using a biopsy needle of at least 16-gauge. Note: RECIST target lesion are not to be biopsied.

I13. Women patient of child-bearing potential must have a negative serum pregnancy test before C1D1 and must agree to use effective forms of contraception from the time of the negative pregnancy test up to 6 months after the last dose of study drugs

I14. Sexually active and fertile men must agree to use contraceptive measures up to 100 days after the last study drugs.

I15. Written informed consent from patient before any study-specific screening procedures, and willingness to comply to study visits and procedures.

I16. Patients must be covered by a medical insurance

Exclusion Criteria:

Non-inclusion 1. Prior exposure to MMD2 inhibitors and/or pazopanib.

Non-inclusion 2. Patients with significant active or uncontrolled cardiovascular disease or prior medical cardiac function disorders including for example uncontrolled hypertension, peripheral vascular disease, congestive heart failure (Class III-IV according to New York Heart Association scale), cardiac arrhythmia, or acute coronary syndrome within 6 months of C1D1 or myocardial infarction, angina pectoris, symptomatic pericarditis, within 12 months of C1D1, congenital long QT syndrome or family history of long QT syndrome and patients with drug eluting stents for cardiovascular purposes.

Non-inclusion 3. Patients diagnosed with treatment-related interstitial lung disease or pneumonitis.

Non-inclusion 4. Patients with secondary malignancy unless this malignancy is not expected to interfere with the evaluation of study endpoints and is approved by the sponsor. Examples of the latter include: basal or squamous cell carcinoma of the skin, in-situ carcinoma of the cervix, localized prostate cancer, prior malignancy and no evidence of disease for ≥ 2 years.

Non-inclusion 5. Patient with any condition (e.g., clinically significant gastrointestinal abnormality or disease resulting in an inability to take oral medication, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow and retain tablets and may affect the absorption of the investigational product are excluded.

Non-inclusion 6. Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:

* Active peptic ulcer disease
* Known intraluminal metastatic lesion(s) with risk of bleeding
* Inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), or other gastrointestinal conditions with increased risk of perforation
* History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment.

Non-inclusion 7. History of hemoptysis, cerebral hemorrhage or clinically significant gastrointestinal (GI) hemorrhage in the past 6 months.

Non-inclusion 8. Hypersensitivity to the active substance or to any of the excipients listed in section VII.1.

Non-inclusion 9. Patients using, or requirement to use while on the study, or not respecting the minimal wash-out period of medications listed below:

Forbidden concomitant medications during the study period and Minimal wash-out period before C1D1:

4 weeks - Any approved anti-cancer treatment (including hormonotherapy, chemotherapy, biological therapy, targeted therapy or immunotherapy) Note: Concurrent use of hormones for non-cancer-related conditions (e.g., insulin for diabetes and hormone replacement therapy) is acceptable. Or Any investigational therapy other than the specified therapies in present protocol

4 weeks - Radiotherapy - Note: Except palliative radiotherapy on non-target lesions after discussion with the Sponsor

4 weeks - Surgery: Major surgical procedure, or significant traumatic injury. Note: If a patient underwent a major surgical procedure, he/she must have adequately recovered from the toxicity (i.e. wound healing) and/or complications from the intervention prior to starting therapy.

4 weeks - Live vaccines. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

1 week - Medicinal products known to prolong the QT interval and/ or to induce "Torsades de Pointes"

1 week - Strong and moderate inducers or inhibitors of CYP3A4/5

1. week - Strong inhibitors of P-glycoprotein (P-gp) or breast cancer resistance protein (BCRP)

   Forbidden concomitant medications during the DLT period:

   unless clinically indicated by institutional and/or American Society of Clinical Oncology (ASCO) guidelines - Growth factors targeting the myeloid lineage
2. weeks prior treatment start and during the DLT defined period - Prophylactic use of red blood cells and platelet transfusions.

Note: Therapeutic transfusions if clinically indicated by institutional and/or ASCO guidelines are permitted but may qualify as DLT. Transfusions outside the above specified timeframe are permitted.

Non-inclusion 10. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis.

Non-inclusion 11. History of (non-infectious) pneumonitis that required steroids, evidence of interstitial lung disease or active non-infectious pneumonitis.

Non-inclusion 12. Known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies) or active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected)

Non-inclusion 13. Pregnant or breast-feeding female patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
for dose escalation part: the Maximum tolerated dose (MTD) of HDM201 given in combination with a fixed dose of pazopanib. | At the end of cycle 2 (each cycle is 21 days)
  The starting dose of HDM201 is 60 mg once every 3 weeks. The dose escalation will be conducted according to a sequential and adaptive Bayesian scheme, using the method of TITE-CRM to determine the MTD of HDM201 in combination with pazopanib.
  The MTD is defined as the dose associated with a probability of Dose Limiting toxicities (DLTs) the closest to 25%. Estimation of MTD will be based upon the estimation of the probability of a DLT.
  DLTs are defined as any of the following adverse events (AE) graded using NCI-CTCAE occurring during the DLT period (2 first cycles) and assessed as related to at least one of the study drugs:
  Grade (G) ≥ 4 neutropenia, G ≥ 3 febrile neutropenia, G ≥ 4 thrombocytopenia or G3 if associated with bleeding and requires platelet transfusion.
  Non-laboratory AEs of G ≥3 for more than 7 days.
  Any G3 or G4 laboratory value if: Medical intervention is required to treat the subjects, or the abnormality leads to hospitalization.
Expansion part: preliminary data on efficacy of the combination in 2 parallel, independent cohorts of Soft-tissue sarcomas according to Murine double minute 2 (MDM2) status: amplified and non-amplified. | 24W
  progression-free rate at 24 weeks (24W-PFR)

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Institut Bergonié, Bordeaux
  - Centre Léon Bérard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No